CLINICAL TRIAL: NCT01039298
Title: Canadian Optically Guided Approach for Oral Lesions Surgical Trial - COOLS
Brief Title: Efficacy of Optically-guided Surgery in the Management of Early-staged Oral Cancer - COOLS TRIAL
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of British Columbia (Other)
Collaborators: Terry Fox Research Institute (Other); British Columbia Cancer Agency (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H09-03090
Record Dates: First submitted 2009-12-22; First posted 2009-12-24 (Estimated); Last update posted 2014-09-10 (Estimated); Status verified 2014-09

CONDITIONS: Oral Cancer; High-grade Precancer
Keywords: Oral cancer; fluorescence visualization; surgical margin; recurrence
MeSH Terms: conditions — Mouth Neoplasms; Margins of Excision; Recurrence

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Active Comparator): All subjects in this study will receive surgery to treat their oral lesions. The margins (or boundaries) of the tissue to be removed during surgery will be defined by 2 different procedures (or study arms) in the operating room.
  The Control arm. Surgical boundaries for oral lesions will be defined under regular white light.
  Interventions: Procedure: Fluorescence visualization device
- B (Experimental): All subjects in this study will receive surgery to treat their oral lesions. The margins (or boundaries) of the tissue to be removed during surgery will be defined by 2 different procedures (or study arms) in the operating room.
  The FV arm (experimental arm). Surgical boundaries for oral lesions will be defined by FV.
  Interventions: Procedure: Fluorescence visualization device

INTERVENTIONS:
Procedure: Fluorescence visualization device — The trial will randomize 200 patients - 100 in the control arm (using conventional white light approach).
  Arms: B
Procedure: Fluorescence visualization device — The trial will randomize 200 patients - 100 in the FV arm (using FV guided the surgery margin)
  Arms: A

SUMMARY:
Oral squamous cell carcinoma (SCC) is a global disease responsible for ~300,000 new cancer cases each year. Local recurrence (~30% of cases) and formation of second primary malignancy are common.2, 3 Cosmetic and/or functional compromise associated with treatment of disease stage is often significant. These statistics underscore the urgent need to develop a better approach in order to control this deadly disease.

It is becoming increasingly apparent that oral cancers develop within wide fields of diseased tissue characterized by genetically altered cells that are widespread across the oral cavity and present in clinically and histologically normal oral mucosa. Complete removal of these lesions is difficult because high-risk changes frequently go beyond clinically visible tumor. In recognition of this, current 'best practice' is to remove SCC with a significant width (usually 10 mm) of surrounding normal-looking oral mucosa. However, since occult disease varies in size such approach often results in over-cutting (causing severe cosmetic and functional morbidity) or under removal of disease tissue, as evidenced by frequent positive surgical margins and high local and regional recurrence - a failure of the 'best practice.

There is a wealth of literature that supports the use of tissue autofluorescence in the screening and diagnosis of precancers in the lung, uterine cervix, skin and oral cavity. This approach is already in clinical use in the lung and the mechanism of action of tissue autofluorescence has been well described in the cervix. Changes in fluorescence reflect a complex interplay of alterations to fluorophores in the tissue and structural changes in tissue morphology, each associated with progression of the disease.

As one of the internationally leading teams in applying tissue fluorescence technology, we have shown that direct fluorescence visualization (FV) tools can identify clinically visible or occult premalignant and malignant lesions that are associated with lesions at risk, with high-grade histology and high-risk molecular change. In a recently small scaled, retrospective study, we have shown that FV helped surgeons in the operating room to determine the extent of the high-risk FV field surrounding the cancer and resulted in remarkably lower 2-year recurrence rates (0% for FV-guided vs. 25% for those without FV-guided approach). There is need to design a larger scale prospective, randomized controlled (Phase III) trial to gather strong evidence in proving the efficacy of the surgery approach using this adjunct tool.

To establish the evidence supporting the change in clinical practice using FV-guided surgery. There are 3 objectives.

2.1. Objective 1 (Clinical evidence): To assess the effect of FV-guided surgery on the recurrence-free survival of histologically confirmed disease within the context of a randomized controlled trial (efficacy). Hypothesis: FV-guided surgery will increase the recurrence-free survival.

2.2. Objective 2 (Quality of Life evidence): To establish the cost per recurrence prevented for this approach and assess quality of life issues. Hypothesis: FV-guided surgery can be delivered in a cost effective manner and improve the quality of life of patients 2.3 Objective 3 (Scientific/Molecular evidence): To assess the presence of previously validated molecular markers (microsatellite analysis, LOH) and histological change (quantitative pathology) in surgical margins in a nested case-control study involving a tumor bank created within this project. Hypothesis: FV-guided surgery will spare normal tissue at the same time improving capture of high-risk tissue.

DETAILED DESCRIPTION:
1.0. OBJECTIVES AND APPROACHES: 1.1. Objective 1 (Clinical evidence): To assess the effect of FV-guided surgery on the recurrence-free survival of histologically confirmed disease within the context of a randomized controlled trial (efficacy).

Hypothesis: FV-guided surgery will increase the recurrence-free survival. Approaches: This Aim requires the establishment of a randomized controlled trial of 200 patients which will compare outcome for patients in 2 arms: one with conventional surgery with margin delineated under white light, and the other using FV guidance for margin delineation. Please see attached Appendix 1 for a step-by-step protocol. This comprises a multidisciplinary team of surgeons, pathologists, project coordinators, and FV Specialists. In addition to the presurgery assessment, all participating patients will have 3-month follow-ups for the first 2 years and 6-month for the rest of the study period. Biopsy will occur when clinically warranted or at 2-year post-surgery.

1.2. Objective 2 (Quality of Life evidence): To establish the cost per recurrence prevented for this approach and assess quality of life issues.

Hypothesis: FV-guided surgery can be delivered in a cost effective manner and improve the quality of life of patients.

Approaches: This aim requires the collection of economic and quality of life (QoL) data to establish the cost per recurrence prevented for FV-guided surgery and to assess quality of life impacts. To asses potential psychosocial consequences of FV-guided surgery we will measure global QoL. We will use the validated EQ-5D and Functional Assessment of Cancer Therapy Head and Neck Module (FACT-H&N) to determine the participant's QoL at each assessment. The questionnaires will be applied at pre-surgery baseline, and at 6-week, 3-month, and 24-month post-surgery follow-ups.

1.3 Objective 3 (Scientific/Molecular evidence): To assess the presence of previously validated molecular markers (microsatellite analysis, LOH) and histological change (quantitative pathology) in surgical margins in a nested case-control study involving a tumor bank created within this project.

Hypothesis: FV-guided surgery will spare normal tissue at the same time improving capture of high-risk tissue.

Approaches: This Aim requires the retrieval and cutting of the archive material for a nested control study. The estimate number of cases reach outcome is 30 (5% of FV group (100) + 25% of control group (100). Additionally, 60 matched controls will be selected (matched by gender, age, smoking habit, and anatomical site). This Aim is critical to demonstrate a shift in field, sparing normal tissue while catching high-risk occult tissue. Samples for the nested molecular analysis will be performed in Rosin's Lab (for microsatellite analysis) and Cancer Imaging at BC Cancer Agency (Dr. MacAulay for qualitative Pathology). The protocols used to analyze these samples have been published.

2.0. STUDY TOOL - VELSCOPE® We have recently developed a simple hand-held field-of-view device for direct visualization of tissue fluorescence in the oral cavity. This tool is currently commercially available as VELScope® (LED Med Inc., White Rock, BC). We have begun a longitudinal study to explore the effect of FV in defining the surgical margin on outcome of oral cancer surgery27. Between 2004 and 2008, 60 patients with a ≤4 cm oral cancer entered the study. Each case was treated with surgical excision alone and was followed for at least 12 months. Thirty-eight patients had FV-guided surgery, with the surgical margin placed at 10 mm beyond the perimeter of autofluorescence loss. The remaining patients (control group) had the surgical margin placed at 10 mm beyond the tumor edge defined by standard white-light examination. Among those, 7 of the 60 cases (12%) have developed a recurrence of severe dysplasia, carcinoma in situ or squamous cell carcinoma at the treated site, all in the control group (25% versus 0%, P = 0.002). These data suggest the potential utility of autofluorescence changes within this clinical setting. There is a need to design a larger scaled randomized controlled clinical trial to confirm the efficacy of FV-guided surgery.

We are also using FV to monitor the potential re-emergence of regions of autofluorescence loss at treated sites in the cases accrued to the longitudinal study and are currently completing an interim assessment of these monitoring results. Autofluorescence loss persists in some cases, increasing in size and intensity over time and giving rise to a clinical lesion containing dysplasia or cancer.

3.0 Core members of the trial and project management We have a well-built core group with long-term and strong working relationships, including surgeons (Drs. Anderson (Co-PI) and Durham), Pathologists (Drs. Berean (Co-PI) and Zhang), and Oral Medicine (Drs. Poh (PI) and Williams), and are in a world-leading position in using fluorescence visualization in operating room and in follow-up. Dr. J. Lee, collaborator, from M.D. Anderson Cancer Centre and has extensive experience in clinical trials with special expertise in randomized controlled trial. He will be the trialist in this project, design a program for patient randomization, oversee the trial protocol, and work with local statistician (Prof. Chen) for day-to-day data management. Professor Jiahua Chen, Department of Statistics, the University of British Columbia will serve as the biostatistician to the trial and will be responsible for the data analysis and submission of interim analyses to the Data Safety Monitoring Board.

4.0 Basic trial design The proposed study will be a double-blinded, randomized controlled Phase III study to evaluate the effect of FV-guided surgery in patients diagnosed with severe dysplasia, carcinoma in situ and invasive squamous cell carcinoma and undergoing surgery treatment with an intent-to-cure. The trial will randomize 200 patients -100 in the FV arm (using FV guided the surgery margin) and 100 in the control arm (using conventional white light approach). The trial period is 5 years - 2 years to complete accrual and 3 more years of follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with severe dysplasia, carcinoma in situ, invasive squamous cell carcinoma (T1 or T2) of the oral cavity (ICO-D site codes: C02.0-C06.9) who will be undergoing curative resection (primary disease).

Exclusion Criteria:

* Patients with a non-oral malignancy diagnosed (not including non-melanoma skin cancer and lymphoma outside of head and neck region) within the past 3 years.
* Patients with evidence of distant metastasis (as determined by CAT and X-ray) at the time of recruitment.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2013-01; Primary Completion 2014-12 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
Recurrence-free survival | 5 years

SECONDARY OUTCOMES:
Histological and molecular evidence of positive margins and quality of life | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Poh, DDS, PhD, Principal Investigator — University of British Columbia; Scott Durham, Dr., Principal Investigator — University of British Columbia; Miriam Rosen, Ph.D, Principal Investigator — Simon Fraser University; Calum MacAulay, Ph.D, Study Director — BC Cancer Agency Research Centre; Penelope Brasher, Ph.D, Study Director — University of British Columbia; Stuart Peacock, Ph.D, Study Director — BC Cancer Agency Research Centre; Kitty Corbett, Ph.D, Study Director — Simon Fraser University; Kenneth Berean, Dr., Study Director — University of British Columbia; Donald Anderson, Dr., Study Chair — University of British Columbia; Michele Williams, DDS, Study Chair — British Columbia Cancer Agency; Joseph Dort, Dr., Study Chair — University of Calgary; Robert Hart, Dr., Study Chair — Dalhousie University; Mike Odell, Dr., Study Chair — University of Ontario; Paul Kerr, Dr., Study Chair — University of Manitoba; John Yoo, Dr., Study Chair — Western University, Canada; Kevin Higgins, Dr., Study Chair — Sunnybrook Hospital; Karen Kost, Dr., Study Chair — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (8):
- Canada (8):
  - University of Calgary, Calgary, Alberta
  - BC Cancer Agency (Vancouver & Fraser Valley Centres) & Vancouver General Hospital, Vancouver, British Columbia
  - CancerCare Manitoba, University of Manitoba, Winnipeg, Manitoba
  - Victoria General Hospital, Dalhousie University, Halifax, Nova Scotia
  - London Health Science Centre, University of Western Ontario, London, Ontario
  - Ottawa General Hospital, University of Ontario, Ottawa, Ontario
  - Sunnybrook Hospital, Toronto, Ontario
  - McGill University Health Centre, Montreal, Quebec

REFERENCES:
- [Derived] Durham JS, Brasher P, Anderson DW, Yoo J, Hart R, Dort JC, Seikaly H, Kerr P, Rosin MP, Poh CF. Effect of Fluorescence Visualization-Guided Surgery on Local Recurrence of Oral Squamous Cell Carcinoma: A Randomized Clinical Trial. JAMA Otolaryngol Head Neck Surg. 2020 Dec 1;146(12):1149-1155. doi: 10.1001/jamaoto.2020.3147. PMID 33034628
- [Derived] Poh CF, Durham JS, Brasher PM, Anderson DW, Berean KW, MacAulay CE, Lee JJ, Rosin MP. Canadian Optically-guided approach for Oral Lesions Surgical (COOLS) trial: study protocol for a randomized controlled trial. BMC Cancer. 2011 Oct 25;11:462. doi: 10.1186/1471-2407-11-462. PMID 22026481